CLINICAL TRIAL: NCT03710889
Title: An Open-Label, Single-Arm, Multicenter Study to Evaluate the Early Effects of Abaloparatide on Tissue-Based Indices of Bone Formation and Resorption
Brief Title: Early Effects of Abaloparatide on Tissue-Based Indices of Bone Formation and Resorption
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA058-05-020
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis; Osteoporosis Vertebral; Osteoporosis Risk; Osteoporosis Fracture; Osteoporosis Localized to Spine; Osteoporosis, Age-Related; Osteoporosis Senile; Osteoporosis of Vertebrae
Keywords: BA058; abaloparatide; TYMLOS®; Bone metabolism; Osteoporosis; Fracture; Bone loss
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Osteoporotic Fractures; Fractures, Bone; Bone Diseases, Metabolic | interventions — abaloparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abaloparatide (Experimental): Participants self-administered a single daily dose of 80 micrograms (µg) of abaloparatide subcutaneously (SC) during the treatment period. Participants were instructed to use a new injection pen after each 30-day period.
  Interventions: Drug: Abaloparatide

INTERVENTIONS:
Drug: Abaloparatide — Abaloparatide is a novel, synthetic, 34 amino acid peptide designed to be a potent and selective activator of the PTH/PTH-related protein (PTHrP) type 1 receptor (PTHR1) signaling pathway with 41% homology to PTH[1-34] and 76% homology to human PTHrP[1-34].
  Other Names: TYMLOS®; BA058

SUMMARY:
The objective of this study is to measure the early effects of abaloparatide on tissue-based bone formation using samples obtained by transiliac crest bone biopsy after quadruple fluorochrome labeling.

DETAILED DESCRIPTION:
This was an open-label, single-arm study of postmenopausal women with osteoporosis treated with 80 micrograms (μg) abaloparatide for 3 months. Transiliac bone biopsies were taken at 3 months after quadruple fluorochrome labeling. The treatment duration of 3 months was determined to be the optimal time when biochemical markers of bone turnover peak and are predictive of subsequent changes in bone mineral density (BMD).

The main study was conducted for a 3-month treatment period with a 1-month follow up. A sub-study was conducted at 1 site to collect peripheral quantitative computed tomography (pQCT) data. Study treatment for participants in the sub-study was extended for an additional 3 months of study drug administration for a total of 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be eligible to participate in this study:

1. The participant is a healthy ambulatory postmenopausal female from 50 to 85 years of age (inclusive) with osteoporosis.
2. The participant has been postmenopausal for at least 5 years. Postmenopausal status will be established by a history of amenorrhea for at least 5 years and by an elevated follicle stimulating hormone (FSH) value of ≥30 international units(IU)/liter (L).
3. The participant has a BMD T-score ≤-2.5 at the lumbar spine (L1-L4) or hip (femoral neck or total hip) by dual-energy x-ray absorptiometry (DXA) or lumbar spine or hip BMD T-score ≤-2.0 with a history of low trauma vertebral, forearm, humerus, sacral, pelvic, hip, femoral, or tibial fracture sustained within 5 years prior to enrollment. These fractures must be documented by radiograph or hospital report.
4. The participant is in good general health as determined by medical history and physical examination (including vital signs), has a body mass index (BMI) of 18.5 to 33, inclusive, and is without evidence of clinically significant abnormality in the opinion of the Investigator.
5. The participant has serum calcium (albumin-corrected), parathyroid hormone (PTH) (1-84), phosphorus, and alkaline phosphatase levels all within the normal range during the Screening Period. Any participant with an elevated alkaline phosphatase value, and who meets all other entry criteria, is required to have a normal bone-specific alkaline phosphatase result to be enrolled.
6. The participant has serum 25-hydroxyvitamin D values ≥ 20 nanograms (ng)/milliliter (mL) and within the normal range. Participants with serum 25-hydroxyvitamin D levels < 20 ng/ml may be treated with vitamin D3 and re-tested once.
7. The participant's resting 12-lead electrocardiogram (ECG) obtained during screening shows no clinically significant abnormality.
8. The participant has read, understood, and signed the written informed consent form.

Exclusion Criteria:

Participants with any of the following characteristics are not eligible to participate in the study:

1. Presence of abnormalities of the lumbar spine that would prohibit assessment of lumbar spine BMD, defined as having at least 2 radiologically evaluable vertebrae within L1-L4.
2. Unevaluable hip BMD or participants who have undergone bilateral hip replacement (unilateral hip replacement is acceptable).
3. History of bone disorders (for example, Paget's disease) other than postmenopausal osteoporosis.
4. Clinically significant abnormality of serum hemoglobin, hematocrit, white blood cells (WBC) and platelets, coagulation, or usual serum chemistry: electrolytes, renal function, liver function and serum proteins.
5. Unexplained elevation of serum alkaline phosphatase.
6. History of radiotherapy (radiation therapy), other than radioiodine.
7. History of bleeding disorder that would preclude a bone biopsy, in the opinion of the Investigator.
8. History of chronic or recurrent renal, hepatic, pulmonary, allergic, cardiovascular, gastrointestinal, endocrine, central nervous system, hematologic or metabolic diseases, or immunologic, emotional and/or psychiatric disturbances to a degree that would interfere with the interpretation of study data or compromise the safety of the participant.
9. History of Cushing's disease, hyperthyroidism, hypo- or hyperparathyroidism, or malabsorptive syndromes within the past year.
10. History of significantly impaired renal function (serum creatinine > 177 micromoles [µmol]/L or >2.0 milligrams [mg]/deciliter [dL]). If the serum creatinine is >1.5 and ≤ 2.0 mg/dL, the calculated creatinine clearance (Cockcroft-Gault) must be ≥ 30 mL/minute (min).
11. History of any cancer within the past 5 years (other than basal cell or squamous cell cancer of the skin).
12. History of osteosarcoma at any time or a history of hereditary disorders which could predispose the participant to osteosarcoma.
13. History of nephrolithiasis or urolithiasis within the past 5 years.
14. Participant known to be positive for hepatitis B, hepatitis C, or human immunodeficiency virus infection (HIV-1 or HIV-2). Testing is not required in the absence of clinical signs and symptoms suggestive of HIV infection or acute or chronic hepatitis.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Radius Health, Inc.
Locations (4):
- United States (4):
  - Panorama Orthopedics & Spine Center, Golden, Colorado
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Harvard Medical School, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hattersley G, Dean T, Corbin BA, Bahar H, Gardella TJ. Binding Selectivity of Abaloparatide for PTH-Type-1-Receptor Conformations and Effects on Downstream Signaling. Endocrinology. 2016 Jan;157(1):141-9. doi: 10.1210/en.2015-1726. Epub 2015 Nov 12. PMID 26562265
- [Background] Cosman F, Miller PD, Williams GC, Hattersley G, Hu MY, Valter I, Fitzpatrick LA, Riis BJ, Christiansen C, Bilezikian JP, Black D. Eighteen Months of Treatment With Subcutaneous Abaloparatide Followed by 6 Months of Treatment With Alendronate in Postmenopausal Women With Osteoporosis: Results of the ACTIVExtend Trial. Mayo Clin Proc. 2017 Feb;92(2):200-210. doi: 10.1016/j.mayocp.2016.10.009. PMID 28160873
- [Derived] Dempster DW, Zhou H, Rao SD, Recknor C, Miller PD, Leder BZ, Annett M, Ominsky MS, Mitlak BH. Early Effects of Abaloparatide on Bone Formation and Resorption Indices in Postmenopausal Women With Osteoporosis. J Bone Miner Res. 2021 Apr;36(4):644-653. doi: 10.1002/jbmr.4243. Epub 2021 Jan 28. PMID 33434314

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abaloparatide
Started | 23
Received at Least 1 Dose of Study Drug (Safety Population) | 23
Bone-Biopsy Population (All enrolled participants who received an evaluable biopsy (defined as a biopsy sample that can be analyzed in the laboratory).) | 19
Completed | 20
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Groups:
- Abaloparatide: Participants self-administered a single daily dose of 80 µg of abaloparatide SC during the treatment period. Participants were instructed to use a new injection pen after each 30-day period.
Arm/Group | Abaloparatide
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
  Other | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram (kg)/square meter (m^2)] | 23.92 (3.629)
Lumbar Spine Bone Mineral Density (BMD) T-Scores [Mean (Standard Deviation); unit: T-Score] — At Baseline, participants were required to have a BMD T-score ≤-2.5 by dual-energy x-ray absorptiometry (DXA) or BMD T-score ≤-2.0 with a history of low trauma vertebral, forearm, humerus, sacral, pelvic, hip, femoral, or tibial fracture sustained within 5 years prior to enrollment. Osteoporosis status was based on the World Health Organization (WHO) 2007 criteria of normal (T-score >-1.0), osteopenia (T-score >-2.5 to ≤-1.0), and osteoporosis (T-score ≤-2.5).
  T-Score
    Total Hip BMD T-Score | -2.392 (0.6363)
    Femoral Neck BMD T-Score | -2.530 (0.5708)
    Lumbar Spine BMD T-Score | -2.232 (1.3098)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mineralizing Surface/Bone Surface (MS/BS) in the Cancellous Envelope at Month 3
Description: Change in dynamic histomorphometry indices was assessed in the cancellous envelope.
Time Frame: Baseline (Day 1), Month 3
Population: The Bone-Biopsy Population included all participants who received an evaluable biopsy (defined as a biopsy sample that can be analyzed in the laboratory). Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of MS/BS
Arm/Group | Abaloparatide
Number analyzed (Participants) | 18
percentage of MS/BS
  Baseline | 5.74 (3.978)
  Change at Month 3 | 18.66 (12.114)
Statistical Analysis 1: Comparison: Abaloparatide; Test type: Other — Within treatment paired t-tests were used to compare the differences in dynamic indices between Baseline and Month 3 using the Bone-Biopsy Population. If the normality assumption is not satisfied at the 0.01 significance level and visual inspection of the data deems it necessary, Wilcoxon signed-rank test is used. No adjustments for multiplicity were made. A 2-sided p-value <0.05 was considered statistically significant; p < 0.0001, Paired t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Bone Formation Rate/Bone Surface (BFR/BS) in the Cancellous Envelope at Month 3
Description: Change in dynamic histomorphometry indices was assessed in the cancellous envelope. BFR/BS was reported as cubic millimeter/square millimeter/year (mm^3/mm^2/year).
Time Frame: Baseline (Day 1), Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3/mm^2/year
Arm/Group | Abaloparatide
Number analyzed (Participants) | 18
mm^3/mm^2/year
  Baseline | 0.011 (0.0076)
  Change at Month 3 | 0.034 (0.0245)

3. Secondary Outcome: Change in Serum Procollagen Type I N-terminal Propeptide (s-P1NP) From Baseline at Month 1 and Month 3
Description: Blood samples were taken to measure efficacy related markers of bone metabolism at Day 1, Month 1, and Month 3.
Time Frame: Baseline (Day 1), Months 1 and 3
Population: The Bone-Biopsy Population included all enrolled participants who received an evaluable biopsy (defined as a biopsy sample that can be analyzed in the laboratory). Here, 'Number Analyzed' signifies participants evaluable for the specified categories.
Measure: Median (Inter-Quartile Range); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Abaloparatide
Number analyzed (Participants) | 19
nanograms (ng)/milliliter (mL)
  Baseline | 54.990 [38.430 to 79.160]
  Change at Month 1: number analyzed (Participants) | 18
  Change at Month 1 | 119.155 [62.810 to 242.240]
  Change at Month 3 | 141.130 [53.420 to 236.980]

4. Secondary Outcome: Change in Serum Carboxy-Terminal Cross-Linking Telopeptide of Type I Collagen (s-CTX) From Baseline at Month 1 and Month 3
Description: Blood samples were taken to measure efficacy-related markers of bone metabolism at Day 1, Month 1, and Month 3.
Time Frame: Baseline (Day 1), Months 1 and 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Abaloparatide
Number analyzed (Participants) | 19
ng/mL
  Baseline | 0.460 [0.308 to 0.549]
  Change at Month 1: number analyzed (Participants) | 18
  Change at Month 1 | 0.052 [-0.109 to 0.174]
  Change at Month 3 | 0.311 [0.079 to 0.694]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Month 4 (main study) and Month 7 (sub-study)
Description: The Safety Population included all enrolled participants who received at least one dose of abaloparatide.
Arm/Group | Abaloparatide
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide (N=23)
Atrial fibrillation (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide (N=23)
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results may not be published prior to the Study Report completion. Investigators may publish results, providing a manuscript to the Sponsor =/> 30 days prior to its submission to a publisher. Sponsor will provide manuscript to Investigators =/> 30 days prior to its submission. Investigator shall comply with Sponsor's policy, withholding publication for an additional 60 days to permit the Sponsor to obtain patent or other proprietary rights protection, if deemed necessary.

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT03710889/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT03710889/SAP_001.pdf